CLINICAL TRIAL: NCT05988476
Title: Investigation of The Efficiency of Pulsed Electromagnetic Field Treatment and Stretching Exercise In Experimental Skeletal Muscle Injury Model
Brief Title: Investıgatıon of The Effıciency of Pulsed Electromagnetıc Field Therapy and Stretching Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mesut ERGAN, Assistant Professor, Suleyman Demirel University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SuleymanDUmesutergan01
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Muscle Injury; Pulsed Electromagnetic Therapy; Muscle Stretching Exercise
Keywords: Muscle Injury; TGF-Beta 1; Fibrosis
MeSH Terms: conditions — Camurati-Engelmann Syndrome; Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention)
- Stretching Exercise (Experimental)
  Interventions: Device: Pulsed Electromagnetic Field Therapy
- Pulsed Electromagnetic Field (Experimental)
  Interventions: Other: Exercise
- Pulsed Electromagnetic Field and Stretching Exercise (Experimental)
  Interventions: Other: Exercise; Device: Pulsed Electromagnetic Field Therapy

INTERVENTIONS:
Other: Exercise — 5 day/week, two week, one session stretching exercises consisting of ten repetitions of one minute
  Arms: Pulsed Electromagnetic Field; Pulsed Electromagnetic Field and Stretching Exercise
Device: Pulsed Electromagnetic Field Therapy — 5 day/week, two week,two sessions consisting of 180 minutes
  Arms: Pulsed Electromagnetic Field and Stretching Exercise; Stretching Exercise

SUMMARY:
In this study, a total of 69 Wistar Albino rats were used, five of which were in the preliminary study. The preliminary study was planned to determine the ideal PEMF treatment time. In the study, animals were divided into 5 groups (Control, INJ, INJ+Exercise, INJ+PEMF, INJ+Exercise+PEMF). Experimental animals were sacrificed on the 7th and 14th days to see the effects of the treatments. At the end of the experiment, genetic, histopathological, and immunohistochemical evaluations were made in the muscle tissue.

DETAILED DESCRIPTION:
Purpose: The aim of this study was to evaluate the efficacy of stretching exercise and the pulsed electromagnetic field (PEMF) method in the treatment of muscle injury (INJ).

Methods: In this study, a total of 69 Wistar Albino rats were used, five of which were in the preliminary study. The preliminary study was planned to determine the ideal PEMF treatment time. In the study, animals were divided into 5 groups (Control, INJ, INJ+Exercise, INJ+PEMF, INJ+Exercise+PEMF). Experimental animals were sacrificed on the 7th and 14th days to see the effects of the treatments. At the end of the experiment, genetic, histopathological, and immunohistochemical evaluations were made in the muscle tissue.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young wistar albino rats

Exclusion Criteria:

* not having any injury

Ages: 10 Months to 11 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Mononuclear cell infiltration, Atrophy and necrosis, Pyknotic nucleus assesment at the end of two weeks | two week
  hematoxylin-eosin staining
VEGF and FGF assesment at the end of two weeks | two week
  immunohischemical staining
TGF-β1, eNOS assesment at the end of two weeks | two week
  Quantitative Reverse-Transcriptase Polymerase Chain Reaction (RT-qPCR)

CONTACTS AND LOCATIONS:
Locations (1):
- SuleymanDU, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No